CLINICAL TRIAL: NCT06601400
Title: Evaluation of Bone Dimensional Changes After Using Xenograft with or Without Erythropoietin Around Immediate Implants in the Esthetic Zone: a Randomized Clinical Trial
Brief Title: Xenograft with or Without Erythropoietin in Immediate Dental Implant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kholoud Sobhy Ibrahim Farag El Deeb, assistant lecturer at future university in egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Erythropoietin,Dental implant
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hopeless Teeth
Keywords: dental implant; Erythropoietin; Xenograft
MeSH Terms: interventions — Erythropoietin; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Test) (Experimental): Immediate implant placement with Xenograft mixed with Erythropoietin
  Interventions: Combination Product: Erythropoietin (EPO) with xenograft
- Group B (Control) (Active Comparator): Immediate implant placement with Xenograft alone
  Interventions: Other: Xenograft alone

INTERVENTIONS:
Combination Product: Erythropoietin (EPO) with xenograft — After atraumatic extraction of the non-restorable tooth, Implant will be placed palatal and apical to osteotomy with at least 2mm gap junction between implant and buccal bone which will be grafted with xenograft and erythropoietin.
  Arms: Group A (Test)
Other: Xenograft alone — After atraumatic extraction of the non-restorable tooth, implant will be placed palatal and apical to osteotomy with at least 2mm gap junction between implant and buccal bone which will be grafted with xenograft alone.
  Arms: Group B (Control)

SUMMARY:
The aim of this study is to evaluate changes in buccal bone thickness after immediate implant placement with xenograft mixed with erythropoietin in the anterior maxilla with a thin buccal bone

DETAILED DESCRIPTION:
PICO:

Population: Patients with non-restorable tooth in anterior maxilla with thin buccal bone (less than 1mm) Intervention: Immediate implant placement with Xenograft mixed with Erythropoietin.

Control: Immediate implant placement with Xenograft alone.

ELIGIBILITY:
* Inclusion criteria

  * Adult (≥18 years) with non-restorable maxillary teeth in the esthetic zone (upper right second premolar to upper left second premolar).
  * Intact with thin labial plate of bone (≤1mm).
  * The recipient site of the implant should be free from any pathological conditions.
  * Patients who are cooperative, motivated and hygiene conscious.
  * Appropriate crown height space to maintain favorable crown : implant ratio
* Exclusion criteria

  * Systemic conditions/diseases that contraindicate surgery.
  * Patients who have any habits that might jeopardize the osseointegration process, such as current smokers.
  * Patients with parafunctional habits that produce overload on implant, such as bruxism and clenching.
  * Patients with periodontal disease.
  * Alcohol or drug abuse.
  * Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-14 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Buccal bone thickness. | 1 year follow up period
  by Cone Beam Computed Tomography (CBCT) in mm

SECONDARY OUTCOMES:
Crestal bone loss | 1 year follow up period
  will be measured by Cone Beam Computed Tomography (CBCT) in mm
Soft tissue thickness. | 1 year follow up period
  will be measured by Endodontic spreader with rubber stopper in mm
The pink esthetic score (PES) | 1 year follow up period
  by taking photographs
Success and survival criteria | 1 year follow up period
  the absence of mobility, the absence of acute or chronic peri-implant infection, the absence of radiolucency around the implant, without pocket probing depth (PPD) ≧ 5 mm, and without vertical bone loss ≧ 1.5 mm in the first year. The cases will be defined as failure if it can't reach any one of the success criteria
Bleeding on probing (BOP) | 1 year follow up period
  According to presence (yes) or absence (No) of bleeding on probing
Pain score | 1, 3, and 7 days
  by using Visual analogue scale from (0-10)
Full-mouth plaque score | 1 year follow up period
  According to presence (yes) or absence(No) of plaque

CONTACTS AND LOCATIONS:
Overall Officials: Noha ghallab, PHD, Study Director — Professor of Oral Medicine and Periodontology, Faculty of Dentistry, Cairo University.; Manar El Zanaty, PHD, Study Chair — lecturer of periodontology
Locations (1):
- Faculty of dentistry, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fettouh AIA, Ghallab NA, Ghaffar KA, Mina NA, Abdelmalak MS, Abdelrahman AAG, Shemais NM. Bone dimensional changes after flapless immediate implant placement with and without bone grafting: Randomized clinical trial. Clin Implant Dent Relat Res. 2023 Apr;25(2):271-283. doi: 10.1111/cid.13178. Epub 2023 Jan 3. PMID 36596471